CLINICAL TRIAL: NCT04809350
Title: Effect of Adjustable Versus Targeted Human Milk Fortification on Weight Gain in Preterm Infants With Birth Weight <1250 g: A Randomized Controlled Trial
Brief Title: Human Milk Fortification With Adjustable Versus Targeted Method
Acronym: FAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REB20-2139
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Growth Failure
Keywords: Human milk; Fortification; Preterm infants
MeSH Terms: conditions — Failure to Thrive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjustable Human Milk Fortification (Active Comparator): Human milk fortification based on blood urea levels
  Interventions: Dietary Supplement: Adjustable Human Milk Fortification
- Targeted Human Milk Fortification (Experimental): Human milk fortification based on milk analysis
  Interventions: Dietary Supplement: Targeted Human Milk Fortification

INTERVENTIONS:
Dietary Supplement: Adjustable Human Milk Fortification — BUN and sodium concentrations will be measured every week in infants on full enteral feeds with fortified human milk.
  Liquid protein will be added based on serum urea.
  Arms: Adjustable Human Milk Fortification
Dietary Supplement: Targeted Human Milk Fortification — Human milk will be analyzed twice weekly. Before the day of analysis, each mother will store fresh milk pumped from 10:00 AM until 8:00 AM of the previous day in a refrigerator and bring it to the hospital.
  Protein, fat, and sodium supplementation will be added to the human milk to meet the recommended daily intakes.
  Arms: Targeted Human Milk Fortification

SUMMARY:
Research question: Do preterm infants born <1250 g achieve better weight gain with targeted fortification compared with the adjustable fortification of human milk?

Hypothesis: Targeted fortification of human milk results in better weight gain in infants with birth weight <1250 gr when compared to the adjustable fortification.

Study design: Open-label, pragmatic, parallel randomized controlled trial in appropriate for gestational age infants with birth weight <1250 g.

DETAILED DESCRIPTION:
Human milk is the ideal diet for neonates. However, it does not provide enough energy, protein, and sodium to meet the nutritional requirements of very preterm infants. Postnatal growth failure is common despite the current use of human milk fortifiers. The main human milk fortification methods include:

1. standard HM fortification (SF) which assumes an average composition of breast milk and adds fortifiers in a fixed dosage. It does not account for variations of nutrient content in human milk
2. Individualized human milk fortification which encompasses two methods:

   1. Adjustable HM fortification (AF): Protein supplementation is provided in addition to SF according to blood urea nitrogen (BUN) concentration which reflects the infant's metabolic response to protein intake. However, there are clinical scenarios in which the BUN levels are not a reliable marker of protein intake, such as acute kidney injury.
   2. Targeted HM fortification (TF): Based on routine analyses of HM that are used to adjust fortification to meet the recommended requirements for infants. It does not take into consideration that the requirements of infants may vary.

SF has frequently failed to achieve appropriate weight gain, while individualized (AF or TF) fortification seems to have better performance. However, the evidence to support one method over the other is lacking.

The objective of the study is to compare weekly average weight gain between preterm infants on AF versus TF.

Once the written consent is obtained, the infant will be randomized to AF or TF. The sequence code will be kept in sequential numbered sealed envelopes. Infants from multiple births will be included as 1 unit and randomized to the same arm of the study.

For patients allocated to the TF group, breast milk will be analyzed twice weekly for energy, protein, and sodium contents. The daily protein, fat, and sodium intakes will be then calculated and optimized to meet the recommended dietary reference intake (DRI) for preterm infants with birth weight <1250 g.

For patients allocated to the AF group, weekly BUN measurements will be performed. Based on BUN concentrations, the liquid protein will be added to achieve the targeted BUN level. Additional calories will be added using formula if growth is suboptimal or DRI is not met based on the assumed human milk content for protein and energy.

The intervention will last 4-8 weeks. For all patients, the day the first BUN concentration and milk analyses are done will be day 1 of intervention. The following measurements will be performed on days 7-8, 14-16, 21-23, and 28-30 of intervention: Weight (grams), length and head circumference (centimeters), BUN and sodium concentrations.

Data on maternal and neonatal characteristics will be collected from their electronic and physical charts.

ELIGIBILITY:
Inclusion Criteria:

* Infants with birth weight <1250 g born at Foothills Medical Centre.
* Appropriate for gestational age (AGA) (according to Fenton's Charts).

Exclusion Criteria:

* Abnormal Newborn Metabolic Screen
* Major congenital anomalies intervention.
* Patients who develop NEC prior to enrollment.
* Patients with confirmed congenital Toxoplasmosis, Syphilis, Rubella, Cytomegalovirus, Herpes simplex virus, Varicella and/or Zika (TORCH infections).
* Patients receiving systemic steroids.
* Patients with acute kidney injury (AKI).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Average weight gain in infants on Adjustable versus Targeted human milk fortification | Weekly for 8 weeks
  Average weight gain measured as g/kg per day

SECONDARY OUTCOMES:
Anthropometrics in infants on Adjustable versus Targeted human milk fortification | Weekly for 8 weeks
  Measurement of head circumference and length in centimeters.
BUN concentration in infants on Adjustable versus Targeted human milk fortification | Weekly for 4 weeks
  mmol/L
Incidence of extra uterine growth restriction | At 36 weeks CA
  Defined as weight less than 10th percentile at 36 weeks corrected age (CA)

CONTACTS AND LOCATIONS:
Overall Officials: Belal Alshaikh, MD, MSc, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada